CLINICAL TRIAL: NCT07215598
Title: Accuracy of Invisalign Attachments: A Split-Mouth Comparative Study of Optimized and Conventional Designs
Brief Title: Split-Mouth Comparison of Invisalign Attachments
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Maria Doughan, Clinical Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00115664
Record Dates: First submitted 2025-10-07; First posted 2025-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Wear, Restoration; Volume Assessment; Clear Aligner Appliance
Keywords: volume assessment; invisalign; clear aligner; digital orthodontics; attachment wear

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized split-mouth (crossover) study evaluating two types of Invisalign attachments: optimized and conventional. Each participant receives both attachment types on contralateral teeth, allowing within-subject comparison of placement accuracy and wear under identical clinical conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Optimized (Active Comparator): Optimized attachments are small, tooth-colored composite bumps placed on teeth during Invisalign treatment to help aligners deliver controlled forces for tooth movement. These attachments are digitally designed in the ClinCheck software to optimize force direction and retention. In this arm, optimized attachments will be bonded according to the manufacturer's standard template and curing protocols. Their bonded geometry and wear over time will be compared to those of conventional attachments placed on the contralateral teeth.
  Interventions: Device: Composite Aligner Attachment
- Conventional (Active Comparator): Conventional attachments are tooth-colored composite bumps placed on teeth during Invisalign treatment to improve aligner retention and control tooth movement. These attachments are designed with standard rectangular or ellipsoid shapes, following established clinical templates. In this arm, conventional attachments will be bonded using manufacturer-recommended materials and curing protocols. Their placement accuracy and wear characteristics will be compared to those of optimized attachments placed on the contralateral teeth within the same participant.
  Interventions: Device: Composite Aligner Attachment

INTERVENTIONS:
Device: Composite Aligner Attachment — Composite aligner attachments are small, tooth-colored resin bumps bonded to specific teeth during Invisalign treatment to enhance aligner retention and force application. These attachments are digitally planned in ClinCheck software and fabricated using manufacturer-provided templates. In this study, two designs: optimized and conventional, will be compared for their accuracy and durability using 3D digital scans at multiple time points.

SUMMARY:
This study evaluates how accurately the attachments used in Invisalign treatment (Align Technology Inc., San Jose, CA, USA) match their planned shapes and sizes in the ClinCheck software (ClinCheck®, Align Technology Inc., San Jose, CA, USA). Attachments are small tooth-colored bumps that help clear aligners grip the teeth and move them effectively.

The investigators are comparing two types of attachments: optimized and conventional, to determine which is bonded to the tooth more accurately and maintains its shape better over time. Participants beginning Invisalign treatment will have attachments placed as part of their normal care. Digital scans will be taken immediately after placement and during follow-up visits to assess attachment accuracy and wear.

The goal is to identify which attachment design provides greater precision and durability to improve the predictability and efficiency of Invisalign treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged18 years or older.
* Patients initiating Invisalign treatment with planned composite attachments.
* Ability to provide written informed consent and agree to additional research intra-oral scans.
* Good oral hygiene and absence of active periodontal disease at enrollment.

Exclusion Criteria:

* Extensive dental restorations (composites, crowns, veneers) on study teeth that could interfere with attachment bonding.
* Enamel defects or severe wear on study tooth surfaces affecting bonding accuracy.
* Contraindications to digital intraoral scanning (e.g., severe gag reflex, metallic prostheses preventing accurate imaging).
* Severe tooth malposition that would compromise accurate attachment placement.
* Poor oral hygiene or active periodontal disease at enrollment and/or if the patient develops poor oral hygiene or active periodontal disease during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Attachment Volume Accuracy | 1 month
  Quantitative comparison of planned versus bonded Invisalign attachment volumes measured using 3D (three dimensional) digital scans. Each bonded attachment will be segmented from intraoral STL (Standard Tessellation Language) files and superimposed onto the corresponding planned ClinCheck model. The absolute difference in attachment volume (in mm³) between planned and bonded models will be calculated to assess bonding accuracy for optimized and conventional designs.
Attachment Active Surface Area Accuracy | 1 month
  Quantitative difference in attachment active surface area using intraoral 3D scans. STL models obtained at baseline (immediately after bonding) and at 1 month will be superimposed to calculate difference in active surface area (mm²). The mean difference between planned and bonded surface areas will be compared for optimized and conventional attachment designs to evaluate bonding precision.
Positional Accuracy | 1 month
  Difference between planned and bonded attachment position, measured as centroid displacement (mm) after 3D registration of STL models at baseline and 1 month.

SECONDARY OUTCOMES:
Volume Reduction Over Time | 6 months
  Quantitative change in attachment volume across follow-up using serial intraoral 3D scans. STL models acquired at baseline (immediately after bonding), 1, 3, and 6 months will be superimposed to calculate absolute loss in attachment volume (mm³) for optimized and conventional designs.
Volume Loss (Percentage) | 6 months
  Relative change in attachment volume expressed as a percentage of the baseline volume. STL models from baseline, 1, 3, and 6 months will be analyzed to calculate mean percent reduction (%) in attachment volume for optimized and conventional designs.
Active Surface Area Change Over Time | 6 months
  Longitudinal change in the active surface area of bonded attachments measured from serial intraoral 3D scans. Segmented STL models at baseline (immediately after bonding), 1, 3, and 6 months will be registered to compute absolute change in active surface area (mm²) for optimized and conventional designs.
Active Surface Area Change (Percentage) | 6 months
  Relative change in attachment active surface area expressed as a percentage of the baseline value. STL models obtained at baseline and at 1, 3, and 6 months will be analyzed to calculate mean percent reduction (%) in active surface area for optimized and conventional attachments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including attachment type, attachment volume, surface deviation, and changes in attachment shape and wear over time, will be shared upon reasonable request. Supporting materials such as the data dictionary, study protocol, statistical analysis plan, informed consent form, and computational methods for volumetric evaluation in MeshMixer will also be made available to qualified researchers for further analysis.
Supporting Information: Study Protocol, SAP
Time Frame: November 2025-July 2028
Access Criteria: De-identified individual participant data (IPD) and supporting documents will be available to qualified researchers upon reasonable request to the Principal Investigator, following approval under the University of Maryland data governance policy.

REFERENCES:
- [Background] Muthuswamy Pandian S, Subramanian AK, Vaiid N. Comparison of efficacy and accuracy of tooth movements in optimized and conventional attachments of clear aligners - A systematic review and meta-analysis. J Oral Biol Craniofac Res. 2025 Sep-Oct;15(5):1123-1133. doi: 10.1016/j.jobcr.2025.07.019. Epub 2025 Jul 29. PMID 40778386
- [Background] Li Q, Yang K. Surface wear of attachments in patients during clear aligner therapy: a prospective clinical study. Prog Orthod. 2024 Feb 19;25(1):7. doi: 10.1186/s40510-023-00506-y. PMID 38369617
- [Background] Fausto da Veiga Jardim A, Curado de Freitas J, Estrela C. Surface wear and adhesive failure of resin attachments used in clear aligner orthodontic treatment. J Orofac Orthop. 2024 May;85(Suppl 1):52-62. doi: 10.1007/s00056-023-00471-5. Epub 2023 Jun 14. PMID 37314488
- [Background] Bellocchio AM, Portelli M, Ciraolo L, Ciancio E, Militi A, Peditto M, Barbera S, Nucera R. Evaluation of the Clinical Variables Affecting Attachment Reproduction Accuracy during Clear Aligner Therapy. Materials (Basel). 2023 Oct 23;16(20):6811. doi: 10.3390/ma16206811. PMID 37895792
- See also: Invisalign Attachments explanation — https://www.invisalign.com/resources/living-with-invisalign/invisalign-attachments